CLINICAL TRIAL: NCT04351074
Title: Ligation of Intersphincteric Track (LIFT) Versus Fistulectomy in Trans-sphincteric Anal Fistula. Randomized Clinical Trial.
Brief Title: Ligation of Intersphincteric Track (LIFT) Versus Fistulectomy in Trans-sphincteric Anal Ffistula.
Acronym: professor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIFT VS fistulectomy
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Transsphincteric Anal Fistula
Keywords: anal fistula, LIFT, fistulectomy
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: group A (39 patients): Patients underwent intersphincteric ligation of fistulous track (LIFT) group B (39 patients): Patients underwent fistulectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A , LIFT (Active Comparator): 39 patients underwnt ligation of the intersphincteric track( LIFT) for treatment of transsphincteric fistula
  Interventions: Procedure: LIFT
- group B fistulectomy (Active Comparator): 39 patients under went fistulectomy for treatment of transsphincteric fistula
  Interventions: Procedure: fistulectomy

INTERVENTIONS:
Procedure: LIFT — ligation of the intersphincteric fistula track
  Arms: group A , LIFT
Procedure: fistulectomy — excision of the fistulous track with its internal and external orifices
  Arms: group B fistulectomy

SUMMARY:
78 patients with transsphincteric fistula allocated into two groups group A underwent LIFT group B u nderwent fistulectomy , comparison between the outcome og both procedures

DETAILED DESCRIPTION:
This randomized comparative clinical trial was carried out in Zagazig university hospitals, general surgery department, between March 2018 and February 2020, on 78 patients with transsphincteric anal fistula.

All patients were informed and signed a written consent for participation in this study, the study was approved by the local ethical committee of our university the sample size was calculated by the statistical unit of the local institutional review board participant selection; participant included in this study are those above 18 years old, suffering transsphincteric anal fistula diagnosed by clinical examination and magnetic resonant imaging (MRI) in doubtful cases, We excluded all patients with;

* Anorectal malignancy.
* Patient with previous radiotherapy to the region.
* Those with fistula due to specific disease as Crohn's disease.
* Patients with anal incontinence.
* Patients with perianal collections.
* Patients on cytotoxic or immunosuppressive therapy. Randomization; According to intervention,participants were randomly allocated using computer generated random numbers into two groups, group A (39 patients): Patients underwent intersphincteric ligation of fistulous track (LIFT) and group B (39 patients): Patients underwent fistulectomy.

Procedures ; All participants were subjected to full clinical examination including detailed history, formal digital rectal examination for assessment of anal sphincter integrity, identification of internal and external openings of the fistula, MRI was performed in those with doubtful clinical examination. Preoperative investigations performed according to American society of anesthesia (ASA) guidelines, all patients received 1 gm third generation cephalosporin with induction of anesthesia and continued for 24 hours postoperative, fleet enema was performed 12 hours and 2 hours before operation.

Surgical technique;

Under spinal anesthesia, participants under went digital rectal examination for identification of the internal and external openings and the fistulous track course, after identification of the external opening it was propped by 14 g cannula through which 2ml hydrogen peroxide was injected and traced through anoscope inside anal canal to identify the internal opening, after that the fistulous track was propped by malleable metal probe, the definitive procedure was then performed according to patient allocation:

in group A; a curvilinear incision was taken in the groove between internal and external anal sphincters over the track course, it was deepened by sharp and blunt dissection between both sphincters till reaching the propped fistulous track, using monopolar diathermy when needed, the track was dissected all around at this point, we used Vicryl 3\0 suture to ligate the fistulous track at two points the medial one as near as possible to the internal sphincter the lateral one is close as possible to the external sphincter, the track was cut in between both ligatures, the lateral part of the track was curetted and the skin around the internal opening was trimmed.

In group B; after identification and probing of the track fistulectomy was carried out by carrying out elliptical incision including internal and external openings, the fistulous track was excised severing the related part of the anal sphincters.

Hemostasis was achieved as needed, wounds was dressed using non adherent dressing, patients received non-steroidal analgesia as per need, patients was discharged after tolerating oral intake.

Follow up; It was achieved via outpatient clinics by the attending surgeon,participants were instructed to attend the clinic every week till complete wound healing , 3 and 6 months after wound healing, later on patients were contacted by phone after 1 year of the procedure, data to be collected throughout follow up included postoperative pain measured by visual analogue scale (VAS) , state of wound healing, state of continence measured by Vaizey score patient's questionnaire, recurrence or persistence of the fistula measured by history and clinical examination.

Statistical analysis; Operative and hospital stay time together with follow up data were collected and statistically analyzed using paired t test and Z test in SPSS program package 22

ELIGIBILITY:
Inclusion Criteria:

* patients with transsphincteric anal fistula

Exclusion Criteria:

* Anorectal malignancy.
* Patient with previous radiotherapy to the region.
* Those with fistula due to specific disease as Crohn's disease.
* Patients with anal incontinence.
* Patients with perianal collections.
* Patients on cytotoxic or immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
recurrence | 8 weeks
  recurrence of the fistula after complete healing of wound detected by clinical examination
incontinence | 1 week
  inability to control flatus or stool detected by Vaizy patient questionnaire
operative time | 1 hour
  time from 1st incision to wound packing counted in minutes
hospital stay | 1 day
  from admission to discharge measured in days
postoperative pain | 1 day
  degree of pain measured by patient questionnaire visual analogue scale(from 1 to 10) the high the score the more sever the pain is

SECONDARY OUTCOMES:
wound complications | 1 week
  bleeding and local wound infection detected by clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: hazem nour, MD, Principal Investigator — zag university
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided